CLINICAL TRIAL: NCT03183973
Title: Effects of Platelet Rich Fibrin (PRF) in Treatment of Non-healing Sternum Wound After Open-heart Surgery
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: SCARM Institute, Tabriz, Iran (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SCARM-Sternum repair
Record Dates: First submitted 2017-05-31; First posted 2017-06-12 (Actual); Last update posted 2020-10-27 (Actual); Status verified 2020-06

CONDITIONS: Sternal Wound Repair

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PRF group (Experimental): patients who will receive Platelet Rich Fibrin (PFR) suspension
  Interventions: Biological: PRF
- placebo group (Experimental)
  Interventions: Biological: placebo group

INTERVENTIONS:
Biological: PRF — patients who will receive PRF suspension
  Arms: PRF group
Biological: placebo group — patients who will receive Placebo
  Arms: placebo group

SUMMARY:
Sternal wound and there complication such as infection, Bruising and scar formation are known as major complication cardiac surgery with a high mortality rate up to 50%. Several approaches have been proposed for treatment of chronic sternal wounds in these patients. however, Underlying confounding factors such as old ages,diabetes mellitus, systemic hypoxia, atherosclerosis and malnutrition have main role against wound repairing. In this study investigators aimed to treatment of patients with open heart surgery and need to strict monitoring of sternal wound repair by Platelet Rich Fibrin.

ELIGIBILITY:
Inclusion Criteria:

* The patient has been diagnosed with an acute STEMI or NSTEMI (confirmed by segment elevation (ST) changes on serial ECG, elevated troponin, coronary artery stenosis or occlusion identified by angiography, and a wall motion abnormality identified by angiography or echocardiography)
* The patient is scheduled to undergo coronary artery bypass surgery.
* The patient does not possess any contraindication for cardiovascular magnetic resonance (CMR).
* The patient is capable of giving informed consent.
* The patient is geographically accessible and willing to return for all follow-up investigations and clinical visits associated with study.

Exclusion Criteria:

* The patient is over the age of 65 years.
* The patient has previous myocardial infarction (MI) (other than the qualifying event) and/or has scar or non-viable myocardium identified by CMR in any other left ventricular (LV) territory.
* The patient is undergoing other cardiac surgery (i.e. concurrent cardiac valve, or aortic surgery).
* The patient requires emergency surgery (i.e. operative intervention (CABG or ventricular assist device) within 24-hrs of assessment).
* The patient has undergone previous cardiac surgery.
* The patient's postsurgical life expectancy is less than 45 days, in the investigator's opinion.
* The patient is of excessively poor baseline health, health-related quality of life, or physical functioning that would preclude a reasonable expected post-operative recovery.
* The patient has received radiotherapy to the chest wall, is receiving immunosuppressive therapy, or is in any way immunocompromised.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2020-03-05 (Actual); Primary Completion 2020-10-15 (Estimated); Study Completion 2020-12-25 (Estimated)

PRIMARY OUTCOMES:
Scar formation | post operative- until release from hospitalization up to 1 month
  Appearance of operative scar diagnose by cardiothoracic surgeon
Wound Infection | post operative- until release from hospitalization up to 1 month
  wound infection incidence diagnose by cardiothoracic surgeon
Bruising | post operative- until release from hospitalization up to 1 month
  Average Bruise Change diagnose by cardiothoracic surgeon

CONTACTS AND LOCATIONS:
Overall Officials: Mohammad Nouri, Ph.D, Study Chair — Head of SCARM Institute; Ahmad Reza Jodati, CTS, Study Director — SCARM institute; Peyman Keyhanvar, MD, Ph.D, Principal Investigator — Deputy for translational medicine of SCARM institute
Locations (1):
- SCARM, Tabriz, East Azarbyjan, Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tashnizi MA, Alamdari DH, Khayami ME, Rahimi HR, Moeinipour A, Amouzeshi A, Seifalian AM. Treatment of non-healing sternum wound after open-heart surgery with allogenic platelet-rich plasma and fibrin glue-preliminary outcomes. Indian J Plast Surg. 2013 Sep;46(3):538-42. doi: 10.4103/0970-0358.122011. PMID 24459346
- [Result] Serraino GF, Dominijanni A, Jiritano F, Rossi M, Cuda A, Caroleo S, Brescia A, Renzulli A. Platelet-rich plasma inside the sternotomy wound reduces the incidence of sternal wound infections. Int Wound J. 2015 Jun;12(3):260-4. doi: 10.1111/iwj.12087. Epub 2013 May 21. PMID 23692143
- [Result] Cotogni P, Barbero C, Rinaldi M. Deep sternal wound infection after cardiac surgery: Evidences and controversies. World J Crit Care Med. 2015 Nov 4;4(4):265-73. doi: 10.5492/wjccm.v4.i4.265. eCollection 2015 Nov 4. PMID 26557476